CLINICAL TRIAL: NCT04211831
Title: An Exploratory Phase 2a Study Evaluating the Efficacy and Safety of URO-902 in Subjects With Overactive Bladder and Urge Urinary Incontinence
Brief Title: URO-902 in Female Subjects With Overactive Bladder and Urge Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: URO-902-2001
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Overactive Bladder With Urge Urinary Incontinence
Keywords: URO-902; hMaxi-K; pVAX/hSlo; Overactive Bladder; Urge Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: URO-902 24 mg; Placebo (Experimental): Participants will receive either a single treatment of URO-902 24 milligrams (mg) or matching placebo.
  Interventions: Drug: URO-902; Drug: Placebo
- Cohort 2: URO-902 48 mg; Placebo (Experimental): Participants will receive either a single treatment of URO-902 48 mg or matching placebo.
  Interventions: Drug: URO-902; Drug: Placebo

INTERVENTIONS:
Drug: URO-902 — intradetrusor injection
  Other Names: hMaxi-K; pVAX/hSlo
Drug: Placebo — intradetrusor injection

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of a single dose of URO-902 24 milligrams (mg) and 48 mg (administered via intradetrusor injection), compared with placebo, in participants with overactive bladder (OAB) and urge urinary incontinence (UUI) up to 48 weeks post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Participant has symptoms of Overactive Bladder (OAB) (frequency and urgency) with Urge Urinary Incontinence (UUI) for a period of at least 6 months prior to screening.
* Participant experiences ≥ 1 episode of UUI per day.
* Participant has not been adequately managed with ≥ 1 oral or transdermal pharmacologic therapies for the treatment of their OAB symptoms.

Exclusion Criteria:

* Participant has symptoms of OAB due to any known neurological reason (e.g., spinal cord injury, multiple sclerosis, cerebrovascular accident, Alzheimer's disease, Parkinson's disease, etc).
* Participant has a predominance of stress incontinence in the opinion of the investigator, determined by participant history.
* Participant currently uses or plans to use medications or therapies to treat symptoms of OAB, including nocturia.
* Participants who have previously been treated with onabotulinumtoxinA for urological indications within 12 months of starting the Screening Bladder Diary, or any other toxin for urological indications, regardless of when treated (participants treated with onabotulinumtoxinA or other toxins for non-urological indications are eligible, regardless of when treated)

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanh Badger, PharmD, Study Director — Urovant Sciences
Locations (20):
- United States (20):
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Orange County Urology Associates, Laguna Hills, California
  - University of Southern California - Norris Hospital, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Stanford University School of Medicine, Palo Alto, California
  - Precision Clinical Research LLC, Sunrise, Florida
  - Iowa Clinic, West Des Moines, Iowa
  - Chesapeake Urology Associates, Hanover, Maryland
  - Bay State Clinical Trials, Watertown, Massachusetts
  - Beaumont Hospital, Royal Oak, Michigan
  - Premier Urology Group, LLC, Edison, New Jersey
  - Urology Center of Englewood, Englewood, New Jersey
  - Great Lakes Physician PC / Western New York Urology Associates, Cheektowaga, New York
  - Accumed Research Associates - ClinEdge - PPDS, Garden City, New York
  - Atrium Healthcare, Charlotte, North Carolina
  - Urology Specialists of The Carolinas, Huntersville, North Carolina
  - Institute For Female Pelvic Medicine, Allentown, Pennsylvania
  - Urology of Virginia, Virginia Beach, Virginia
  - Washington Urology & Urogynecology Associates, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, randomized, double-blind, placebo-controlled, single-treatment, 2-cohort, dose escalation study evaluated the efficacy and safety of URO-902 in females with overactive bladder (OAB) and Urge Urinary Incontinence (UUI).
Pre-assignment Details: A total of 80 participants were randomized into the study.
Groups:
- Placebo: Participants were sequentially randomized in a 2:1 ratio to receive either URO-902 24 milligrams (mg) or placebo as a single treatment, administered by intra-detrusor injections via cystoscopy.
- URO-902 24 mg: Participants were sequentially randomized in a 2:1 ratio to receive either URO-902 24 mg or placebo as a single treatment, administered by intra-detrusor injections via cystoscopy.
- URO-902 48 mg: Participants were sequentially randomized in a 2:1 ratio to receive either URO-902 48 mg or placebo as a single treatment, administered by intra-detrusor injections via cystoscopy.
Period: Overall Study
Arm/Group | Placebo | URO-902 24 mg | URO-902 48 mg
Started | 27 | 26 | 27
Completed | 23 | 22 | 22
Not Completed | 4 | 4 | 5
Not completed — Withdrawal by Subject | 4 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Unable to Complete the Procedures Successfully | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent- to-treat Exposed (ITT-E) population was defined as all participants who were randomized and treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | URO-902 24 mg | URO-902 48 mg | Total
Number analyzed (Participants) | 26 | 22 | 26 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (7.05) | 65.7 (7.39) | 62.8 (6.75) | 64.7 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 26 | 74
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 1 | 7
  Not Hispanic or Latino | 24 | 18 | 25 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 7 | 17
  White | 20 | 17 | 19 | 56
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 12 in Average Daily Number of Urgency Episodes
Description: Average daily number of urgency episodes was calculated as the total number of urgency episodes recorded on a completed diary day within the visit window divided by the number of days the Bladder Diary was filled out. An urgency episode was defined as when a participant answered "Yes" to the question "Need to urinate immediately" on the bladder diary electronic case report form (eCRF). If a participant had more than 1 bladder diary filled out on the same day, then all the urgency episodes were summed together. The denominator used for calculating the average number only counted the days in which there was at least 1 completed bladder diary day within the visit window. Baseline was defined as the last non-missing measurement prior to the study treatment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and at Week 12
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Urgency episodes per day
Arm/Group | Placebo | URO-902 24 mg | URO-902 48 mg
Number analyzed (Participants) | 21 | 22 | 21
Urgency episodes per day | -1.13 (0.740) | -2.43 (0.777) | -3.37 (0.738)
Statistical Analysis 1: Comparison: Placebo vs URO-902 24 mg; Test type: Other; p = 0.1722, mixed model for repeated measures; Least square mean difference = -1.29, 95% CI 2-sided [-3.16 to 0.58] — Treatment comparison between Placebo and URO-902 24 mg using least sqaure mean difference and 95% confidence interval (CI) has been presented
Statistical Analysis 2: Comparison: Placebo vs URO-902 48 mg; Test type: Other; p = 0.0159, Mixed model for repeated measures; Least Square Mean Difference = -2.24, 95% CI 2-sided [-4.04 to -0.43] — Treatment comparison between Placebo and URO-902 48 mg using least sqaure mean difference and 95% CI has been presented

2. Secondary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant, administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize participant and may require medical or surgical intervention to prevent any of outcomes listed above. TEAEs/TESAEs are defined as any event that began or worsened in severity after initial exposure of study treatment through 48 weeks after treatment administration or the date of the initiation of another overactive bladder medication, investigational agent, or surgical intervention, whichever occurred first.
Time Frame: Up to Week 48
Population: Safety Population comprises of all participants who were randomized and received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | URO-902 24 mg | URO-902 48 mg
Number analyzed (Participants) | 26 | 22 | 26
Participants
  Any TEAE | 14 | 10 | 14
  Any TESAE | 3 | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 48 Weeks
Description: Treatment emergent adverse events (TEAEs) and Treatment emergent serious adverse events (TESAEs) were collected in Safety Population. Safety Population comprised of all participants who were randomized and received study drug.
Arm/Group | Placebo | URO-902 24 mg | URO-902 48 mg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22 | 0/26
Serious Adverse Events (participants affected / at risk) | 3/26 | 1/22 | 2/26
Other Adverse Events (participants affected / at risk) | 14/26 | 10/22 | 14/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | URO-902 24 mg (N=22) | URO-902 48 mg (N=26)
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (General disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | URO-902 24 mg (N=22) | URO-902 48 mg (N=26)
Urinary tract infection (Infections and infestations) | 1 | 0 | 4
Bacteriuria (Infections and infestations) | 0 | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 2
Device intolerance (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Suprapubic pain (General disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
ECG signs of myocardial infarction (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1
Residual urine volume increased (Investigations) | 0 | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor does not object to publication by Institution or Principal Investigator (PI) of results of the Trial based on information collected or generated by the Institution or PI. However, the Institution and PI are required to provide the Sponsor with an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed to ensure against any inadvertent disclosure of Sponsor Confidential Information or unprotected Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT04211831/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT04211831/SAP_001.pdf